CLINICAL TRIAL: NCT04165837
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral FB-101 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Oral FB-101 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 1ST Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1ST-102-01
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: FB-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB-101 — Part A - Single Ascending Dose study Part B - Multiple Ascending Dose study
  Arms: Active
Drug: Placebo — Part A - Single Ascending Dose matching placebo study Part B - Multiple Ascending Dose matching placebo study
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of oral doses of FB-101 in healthy subjects.

DETAILED DESCRIPTION:
Part A

* To assess the safety and tolerability of single ascending oral doses of FB-101 in healthy subjects.
* To assess the pharmacokinetics (PK) of single ascending oral doses of FB-101 in healthy subjects.
* To assess the effect of a high-fat meal on the PK of a single oral dose of FB-101 when administered to healthy subjects.

Part B

* To assess the safety and tolerability of multiple ascending oral doses FB-101 in healthy subjects.
* To assess the PK of multiple ascending oral doses of FB-101 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non childbearing potential only) 19 55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to (the first) dosing and throughout the study, based on subject self reporting.
3. Body mass index (BMI) ≥ 18 and ≤ 32.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, neurological examination, ophthalmic examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. A female subject must be of non childbearing potential and must have undergone one of the following sterilization procedures at least 6 months prior to (the first) dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or
   * be postmenopausal with amenorrhea for at least 1 year prior to (the first) dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after (the last) dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to (the first) dosing of study drug. A male who has been vasectomized less than 4 months prior to study (first) dosing must follow the same restrictions as a non vasectomized male).
7. If male, must agree not to donate sperm from the first dosing until 90 days after (the last) dosing.
8. Able to swallow multiple capsules.
9. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

* 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.

  2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.

  3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

  4. Is at suicidal risk in the opinion of the PI as per the following criteria:
  1. Any suicide attempts within 12 months prior to screening or any suicidal intent, including a plan, within 3 months prior to screening.
  2. C-SSRS answer of "YES" on suicidal ideation within 3 months prior to screening. 5. History or presence of alcoholism or drug abuse within the past 2 years prior to (the first) dosing.

     6. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.

     7. History of allergy to lignocaine/fluorescein (LF) or tropicamide (T) (eye examination agents).

     8. History of seizures (childhood febrile seizures are excepted). 9. Female subjects of childbearing potential. 10. Female subjects with a positive pregnancy test or who are lactating. 11. Positive urine drug or alcohol results at screening or check in. 12. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).

     13. Supine blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.

     14. Supine heart rate is lower than 40 bpm or higher than 99 bpm at screening. 15. Estimated creatinine clearance <90 mL/min at screening. 16. Unable to refrain from or anticipates the use of any drug including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study. Drugs known to be significant inducers of cytochrome P450 (CYP) enzymes and/or P-glycoprotein (P gp), including St. John's Wort will be prohibited for 28 days prior to the first dosing and throughout the study. After dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee. For subjects having CSF sampling, topical medication for minor dermatological conditions, stool softeners, local anesthetics, and/or intravenous normal saline may be permitted as appropriate for lumbar puncture procedure for CSF sample collection at the discretion of the PI.

     17. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to (the first) dosing and throughout the study.

     18. Donation of blood or significant blood loss within 56 days prior to (the first) dosing.

     19. Plasma donation within 7 days prior to (the first) dosing. 20. Participation in another clinical study within 30 days prior to the (first) dosing. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 (of Period 1 for the Fed Cohort) of the current study.

     21. History or presence of: risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome); sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities.

     22. Has an abnormal screening ECG indicating a second- or third- degree AV block, or one or more of the following: QRS > 120 msec, QTcF > 450 msec for males and > 460 msec for females, PR interval > 220 msec. Any rhythm other than normal sinus rhythm, which is interpreted by the PI or designee to be clinically significant at screening or check-in.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment emergent adverse events (TEAEs) | 7 days after the last dose
  To assess the safety and tolerability of single and multiple ascending oral doses of FB-101 in healthy adult subjects

SECONDARY OUTCOMES:
Peak plasma concentration of FB-101 in plasma | 72 hours after the last dose
  PK of FB-101
Area under the plasma concentration versus time curve of FB-101 in plasma | 72 hours after the last dose
  PK of FB-101
Peak plasma concentration of FB-101 in plasma under fed condition | 72 hours after the last dose
  Food effect on the PK of FB-101
Area under the plasma concentration versus time curve of FB-101 in plasma under fed condition | 72 hours after the last dose
  Food effect on the PK of FB-101

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL, Baltimore, Maryland, United States